CLINICAL TRIAL: NCT02311153
Title: Safety and Efficacy of Laryngeal Mask Airways in Sinonasal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Justin Turner, Assistant Professor of Otolaryngology-Head and Neck Surgery, Assistant Professor of Biomedical Engineering, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 141421
Record Dates: First submitted 2014-11-10; First posted 2014-12-08 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Conditions Requiring Sinonasal Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endotracheal intubation (Active Comparator): Endotracheal intubation for airway management and ventilation during sinonasal surgical procedure
  Interventions: Device: Mallinckrodt Endotracheal Tube (ETT)
- Laryngeal mask airway (Experimental): Laryngeal mask for airway management and ventilation during sinonasal surgical procedure
  Interventions: Device: Laryseal Laryngeal mask airway (LMA)

INTERVENTIONS:
Device: Mallinckrodt Endotracheal Tube (ETT) — Patient is intubated for airway protection and ventilation with the Mallinckrodt ETT.
  Arms: Endotracheal intubation
Device: Laryseal Laryngeal mask airway (LMA) — Laryseal Laryngeal mask airway is used to provide airway protection and ventilation.
  Arms: Laryngeal mask airway

SUMMARY:
Laryngeal mask airways (LMA) have been shown to be a safe mode of airway management when delivering general anesthesia to patients during a variety of operative procedures. LMA's have been studied in a wide range of otolaryngologic procedures, and are generally safe and accepted by both anesthesia providers and surgeons alike. This study will aim to demonstrate the safety and efficacy of LMA for airway management during sinonasal surgery by directly comparing them to endotracheal intubation in a prospective randomized single-blind study.

DETAILED DESCRIPTION:
LMA's have been studied in a wide range of otolaryngologic procedures, and are generally safe and accepted by both anesthesia providers and surgeons alike, as a safe mode of airway management when delivering general anesthesia. In sinonasal surgery, however, there are more concerns regarding the use of LMA's for airway management. Due to the nature of sinonasal procedures, the patient is exposed to blood and secretions that may drip/flow from the nasal cavity into the oropharynx and potentially into the upper and lower airways if not protected adequately. Additionally, often times, manipulation of the patient's head throughout the procedure is encountered to improve operative positioning. As a result, both surgeons and anesthesiologists have been hesitant to utilize LMA's in these types of surgeries despite documented benefits of increased patient comfort, fewer hemodynamic fluctuations during induction of anesthesia, and better controlled emergence when using LMA's.

Specific Aims The overall purpose of this study is to demonstrate the ability to provide safe and effective ventilation and airway protection with a laryngeal mask airway (LMA) during sinonasal surgery, by directly comparing them to endotracheal intubation in a prospective randomized single-blind study.

Aim 1: Analyze and compare the incidence and severity of airway contamination/aspiration of blood and secretions during sinonasal surgery and reveal any statistically significant difference between LMA and endotracheal intubation.

Aim 2: Analyze and compare the incidence of various outcome measures including laryngospasm, bronchospasm, anesthesia time, recovery time, post-op pain medication requirements, and airway complications between LMA and endotracheal intubation.

Aim 3: Analyze and compare both patient comfort and surgeon satisfaction after procedure between LMA and endotracheal intubation groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 yo or older) undergoing elective sinonasal procedures including rhinoplasty, septoplasty, and paranasal sinus surgery estimated blood loss will be less than 300cc and the length of the procedure will be expected to last 2 hours or less
* American Society of Anesthesiologists (ASA) scores 1-3
* Mallampati classification 1-3

Exclusion Criteria:

* Currently pregnant
* History of obstructive sleep apnea with history of difficulty with ventilation
* Mouth opening less than 3cm
* Indications for fiberoptic intubation present
* Upper aerodigestive tract mass or malignancy
* Procedure deemed emergent
* Severe gastroesophageal reflux, severe cardiac, pulmonary, renal or hepatic co-morbidities
* Unable to consent to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Turner, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was completed in clinic and the pre-operative surgical area.
Pre-assignment Details: 2 patients were consented and enrolled in the clinic setting, but they did not end up being randomized:
  1 did not proceed with surgery
  1 was diagnosed with sleep apnea, which is exclusionary
Period: Overall Study
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Started | 53 | 49
Completed | 48 | 42
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway | Total
Number analyzed (Participants) | 53 | 49 | 102
Age, Categorical [Count of Participants; unit: Participants] — Date of birth was collected from the medical record and confirmed at date of surgery.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 35 | 45 | 80
    >=65 years | 18 | 4 | 22
Sex: Female, Male [Count of Participants; unit: Participants] — Sex was recorded from the medical record, with in-person confirmation at clinic visit(s).
  Participants
    Female | 25 | 29 | 54
    Male | 28 | 20 | 48
Region of Enrollment [Number; unit: participants]
  United States | 53 | 49 | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Presence or Absence of Blood/Secretions in Trachea and Larynx Based on Soiling Score
Description: Presence or absence of blood/secretions as noted in trachea and larynx. Patients were evaluated based on a soiling score completed by the surgeon, ranging from 0 (no contamination or soilage) to 3 (contamination of the tube/bloody secretions).
Time Frame: intraoperative, within about 1 hour
Population: Participants that started the study were analyzed. Data was missing for 1 participant in each arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 52 | 48
Participants
  Soilage score 0 | 12 | 10
  Soilage score 1 | 15 | 21
  Soilage score 2 | 15 | 10
  Soilage score 3 | 10 | 7

2. Secondary Outcome: Anesthesia Time in Minutes
Description: Start and stop time of anesthesia as recorded in anesthesia record
Time Frame: beginning and end of anesthesia (approximately 2 hours)
Measure: Mean (Full Range); unit: minutes
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 53 | 49
minutes | 61 [11 to 167] | 49 [17 to 156]

3. Secondary Outcome: Recovery Time in Minutes
Description: Minutes spent in recovery room as recorded in the recovery room record
Time Frame: time spent in recovery room after surgery (approximately 4 hours)
Population: Participants that started the study were analyzed.
Measure: Mean (Full Range); unit: minutes
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 53 | 49
minutes
  PACU phase 1 time | 34.5 [7 to 111] | 30 [5 to 112]
  PACU phase 2 time | 37.5 [2 to 181] | 40 [0 to 220]

4. Secondary Outcome: Presence of Laryngeal Spasm
Description: As recorded in anesthesia care record
Time Frame: From start of anesthesia through hospital discharge (approximately 6 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 53 | 49
Participants | 0 | 0

5. Secondary Outcome: Post-op Pain Med Requirements
Description: Recording pain medications given to patient as noted in the recovery room records and medication administration record
Time Frame: 48 hour medicine requirement
Population: Participants that started the study were analyzed. Data was missing for 5 participants in the Endotracheal intubation arm and 7 participants in the Laryngeal mask airway arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 48 | 42
Participants
  > 15 pills | 0 | 0
  10-14 pills | 2 | 3
  5-9 pills | 3 | 8
  1-4 pills | 21 | 13
  No pain meds taken | 22 | 18

6. Secondary Outcome: Presence or Absence of Airway Complications
Time Frame: Start of surgery through hospital discharge (approximately 6 hours)
Population: Participants that started the study were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 53 | 49
Participants
  Presence of airway complications | 0 | 0
  Absence of airway complicaitons | 53 | 49

ADVERSE EVENTS:
Time Frame: Patients are monitored for adverse events from the start of surgery through hospital discharge (approximately 6 hours) and are contacted again at first post-op visit, about 5 to 7 days later.
Description: Throughout the surgical procedure, the patient is monitored for any adverse events including desaturation of oxygen saturation, the occurrence of bronchospasm, laryngospasm, and other airway complications.
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/49
Other Adverse Events (participants affected / at risk) | 0/53 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes